CLINICAL TRIAL: NCT01918046
Title: MIOX for Early Detection of Acute Kidney Injury After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Barnes-Jewish Hospital (Other)
Responsible Party: Principal Investigator, Anitha Vijayan, MD, Professor of Medicine, Washington University School of Medicine
Other Study IDs: MIOX-1
Record Dates: First submitted 2013-07-30; First posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Acute Kidney Injury
Keywords: biomarker; MIOX
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Only for analysis of biomarker
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a single-center, prospective sample collection study. Samples will be used to establish the performance characteristics of myo-inositol oxygenase (MIOX) as an aid in the early diagnosis of acute renal injury (AKI) following cardiac surgery.

DETAILED DESCRIPTION:
Approximately 100 adults scheduled to undergo cardiac surgery involving the use of cardiopulmonary bypass will be eligible for enrollment in this study. Blood and urine samples will be obtained from all patients in the study for future measurement of both MIOX and creatinine concentrations in the same sample at each of the following time points:

* Baseline (within 24 hours prior to the start of surgery)
* Immediately following cardiopulmonary bypass (time 0), 3 (± 1), 6 (± 2), 12 (+/-2) 18 (± 2), and 24 (± 2) hours following cardiopulmonary bypass.

Urine and lithium heparin anti-coagulated blood will be collected at each time point. Blood and urine samples will be immediately centrifuged, aliquoted, and frozen at -80oC prior to analysis. Samples will be stored and analyzed at Washington University School of Medicine.

The results of these assessments will be blinded to the medical team during the study and will not impact the medical management of the patient.

Serum creatinine measurements obtained by the medical team as part of routine care both pre-operatively and post-operatively as well as any additional post-operative renal insults, the development of oliguria, need for a nephrology consultation, length of intensive care unit (ICU) stay, initiation of dialysis and mortality will be recorded through Day 10. Patients will be followed throughout their hospital stay, which on average is expected to be about 10 days.

The statistical analysis will evaluate the correlation of plasma and urine MIOX (absolute and change from baseline) with parameters indicative of renal injury (e.g., increases in plasma creatinine through Day 5 and development of oliguria, need for a nephrology consult or initiation of dialysis through Day 10). These results will assist in establishing the sensitivity and specificity of plasma and urine MIOX for the detection of meaningful kidney injury following cardiopulmonary bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female scheduled for cardiac surgery including placement of Left or Right ventricular assist devices, requiring cardiopulmonary bypass
2. Age greater than or equal to 18 years

Exclusion Criteria:

1. Age less than 18 years
2. Inability to obtain Informed Consent from patient or representative
3. Prisoners or other institutionalized or vulnerable individuals.
4. Participation in an interventional clinical study within the previous 30 days.
5. History of previous renal transplantation
6. Stage 4 or 5 chronic kidney disease (estimated GFR< 30 mL/min/1.73m2)
7. Known or suspected ongoing pre-operative acute renal failure due to any cause, including pre-renal, intrinsic renal or post-renal (obstructive) etiologies (as evidenced by increasing serum creatinine or oliguria pre-operatively)
8. Already receiving dialysis, in imminent need of dialysis or considered highly likely to need dialysis in the immediate post-operative period for fluid management.
9. Any known or suspected renal ischemic or nephrotoxic insult (such as cardiac arrest, intravenous contrast procedure, etc) during the 48 hrs prior to surgery.
10. Known or suspected infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV) infection; hepatitis B virus (HBV) infection or other infectious hepatitis.
11. Pre-operative hematocrit < 25%, recent blood transfusions have been administered to maintain hematocrit > 25% or any other contraindication to obtaining the study specified blood samples.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery at BJH
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury | 10 days

SECONDARY OUTCOMES:
Renal replacement therapy | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Gaut, MD, PhD, Principal Investigator — Washington University School of Medicine; Anitha Vijayan, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States